CLINICAL TRIAL: NCT04645004
Title: Impact of Maternal Aspirin Tehrapy on the Maternal/Fetal Unit at Delivery: a Study of Aspirin Pharmacokinetics, Pharmacodynamics, and Pharmacogenomics Through Pregnancy
Brief Title: Antenatal Platelet Response on Aspirin: a Pharmacokinetic Study Through Pregnancy
Acronym: APROACH-PK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); March of Dimes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20F.911; 3R21HD101127-01S1 (NIH)
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: One arm PK/PD study of aspirin in pregnancy1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Aspirin (Other): 81mg aspirin daily
  Interventions: Drug: Aspirin 81Mg Non-enteric coated Tab

INTERVENTIONS:
Drug: Aspirin 81Mg Non-enteric coated Tab — one tab daily

SUMMARY:
Longitudinal pharmacokinetic and pharmacodynamic study in first and third trimester of pregnancy

DETAILED DESCRIPTION:
This will be a longitudinal addition to an existing R21cohort enrolled in the first trimester to include a first and third trimester assessment of pharmacokinetics/pharmacodynamics (PK/PD) of aspirin and how individual factors impact aspirin PK/PD in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* <16 weeks' gestational age
* Singleton pregnancy
* Plan to take 81mg aspirin due to high risk history (below), but not yet initiated
* ≥1 risk factor:

  * Chronic hypertension
  * Type I or II diabetes
  * Previous preeclampsia
  * Renal disease
  * Autoimmune disease (SLE) OR

    ≥2 risk factor:
  * Nulliparity
  * IVF pregnancy
  * Black race or socioeconomic disadvantaged
  * BMI>30
  * Prior adverse pregnancy outcome

Exclusion Criteria:

* Contraindication to aspirin
* Current or planned use of any other anticoagulation
* Current need for dialysis
* Use of aspirin therapy prior to enrollment in the current pregnancy
* Thrombocytopenia (<150)
* Other known platelet disorder/thrombophilia at enrollment

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
salicylic acid level | 24 hour
  time/concentration profile
serum thromboxane | 4 week post initiation
  ELISA based quantification of serum thromboxane B2
PFA-100 | 4 week post initiation
  PFA-100 epi closure time (Siemens)

SECONDARY OUTCOMES:
Urinary thromboxane | 4 week post initiation
  ELISA based quantification of urindary dehydrothromboxane B2

CONTACTS AND LOCATIONS:
Overall Officials: Rupsa C Boelig, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final results of this study will plan to be submitted for publication within 12 months of completion of analysis of samples. Following publication, a data set excluding any protected health information will be available on request pending agreement on use of data and appropriate IRB approval for data sharing agreement with the outside individuals or institutions requesting data. The data sharing agreement will provide that the individual/institution requesting the data will commit to using the data only for research purposes and not attempt to identify any individual participant, to secure the data using appropriate computer technology and security, and finally to destroy or return the data set after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Following publication of data, 12 months following study completion
Access Criteria: The data sharing agreement will provide that the individual/institution requesting the data will commit to using the data only for research purposes and not attempt to identify any individual participant, to secure the data using appropriate computer technology and security, and finally to destroy or return the data set after analyses are completed.